CLINICAL TRIAL: NCT02195791
Title: Mechanism of Hyperglycemia and Neuroprotection Effect of Pioglitazone in Acute Ischemic Stroke
Brief Title: Neuroprotection of Pioglitazone in Acute Ischemic Stroke
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Diffculty in participant enrollment
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOHW103-TDU-B-212-113001 S
Record Dates: First submitted 2014-07-14; First posted 2014-07-21 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone (Active Comparator)
  Interventions: Drug: Pioglitazone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone 30mg/tab (oral) 1 tab once daily for 7 days
  Arms: Pioglitazone
Drug: Placebo — Placebo (oral) 1 tab once daily for 7 days
  Arms: Placebo

SUMMARY:
Pioglitzone, an oral anti-diabetic drug which can reduce insulin resistance and decrease inflammation. It has been proven to be an effective neuroprotective agent in animal model of ischemic stroke. In this study, the investigators will conduct a phase II clinical trial (double-blind, randomized placebo controlled study) to survey the neuroprotection effect of pioglitazone in stroke patients with hyperglycemia. A total of 152 acute ischemic stroke patients with hyperglycemic will receive insulin or sulfonyurea for blood sugar control, and will be randomly randomized into intervention (Pioglitazone 30mg once a day p.o,) and control group (placebo). The investigators expect to prove the neuroprotective efficacy of Pioglitazone in acute stroke with hyperglycemia and identify the biomarkers associated with good neurological outcome in patients with Pioglitazone treatment from the investigators clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke onset within 48 hours
2. Age≧20 years
3. Stroke severity with at least one point for limb weakness in National Institutes of Health Stroke Scale (NIHSS).
4. The patients with no known history of diabetes with admission serum glucose ≧130 mg/dl.

Exclusion Criteria:

1. The patients who have history of urinary bladder cancer or hematuira.
2. The patients who have history of congestive heart failure or myocardial infarction.
3. The patients who have known history of using pioglitazone before the onset of stroke.
4. The patients who have mRS≧3 before stroke onset.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) | Day 90 after stroke

SECONDARY OUTCOMES:
National Institute of Health Stroke Scale (NIHSS) | Day 90 after stroke
Barthel's Index | Day 90 after stroke

CONTACTS AND LOCATIONS:
Overall Officials: Nai-Fang Chi, MD, Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Taipei Medical Universtiy- Shuang Ho Hospital, New Taipei City, Taiwan